CLINICAL TRIAL: NCT05462392
Title: Robot-assisted Urological Surgeries Using the MicroHand S Robot: a Prospective, Single Blind, Randomized Controlled Trial
Brief Title: Robot-assisted Urological Surgeries Using the MicroHand S Robot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NKJSSQXCKXT02-WG
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer; Prostate Cancer; Renal Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Micro Hand S robot group (Experimental): 68 patients were randomly allocated in the Micro Hand S robot group and partial nephrectomy, radical cystectomy, and radical prostatectomy will be performed using the Micro Hand S robot.
  Interventions: Device: robot-assisted surgery
- the da Vinci robot group (Other): 68 patients were randomly allocated in the da Vinci robot group and partial nephrectomy, radical cystectomy, and radical prostatectomy will be performed using the da Vinci robot.
  Interventions: Device: robot-assisted surgery

INTERVENTIONS:
Device: robot-assisted surgery — urological surgeries, such as partial nephrectomy, radical cystectomy, and radical prostatectomy was performed for patients using the Micro Hand S robot group.
  Arms: the Micro Hand S robot group
Device: robot-assisted surgery — urological surgeries, such as partial nephrectomy, radical cystectomy, and radical prostatectomy was performed for patients using the da Vinci robot group
  Arms: the da Vinci robot group

SUMMARY:
A single-blinded, prospective randomized parallel controlled clinical trial is designed and will be conducted from July 2022 to November 2023 (anticipated). One hundred and thirty-six patients (anticipated) with renal cancer or bladder cancer or prostate cancer will be enrolled in this study. Those patients will be enrolled by two hospital centers and the patients will be randomly divided into the Micro Hand S surgical robot group and the da Vinci surgical robot group. Robot-assisted partial nephrectomy, radical cystectomy, and radical prostatectomy will be conducted using the Micro Hand S robot or the da Vinci robot. The success rate of operation, assembly time, operation time, intraoperative hemorrhage, continence rate (if applicable), postoperative pain, comprehensive complication index, resident time and surgeon satisfaction were recorded. The aim of the study is to determine whether the newly developed Chinese Micro Hand S surgical robot results in non-inferiority outcomes in urological surgeries compared with the prevalent da Vinci robot.

DETAILED DESCRIPTION:
Objective: To determine whether the newly developed Chinese Micro Hand S surgical robot results in non-inferiority outcomes in partial nephrectomy, radical cystectomy, and radical prostatectomy, compared with the prevalent da Vinci robot.

Design: A single-blinded, prospective randomized parallel controlled clinical trial will be conducted from July 2022 to November 2023 (anticipated). One hundred and thirty-six patients (anticipated) with renal cancer or bladder cancer or prostate cancer will be enrolled in this study. Those patients will be enrolled by two hospital centers and the patients will be randomly divided into the Micro Hand S surgical robot group and the da Vinci surgical robot group.

Interventions: Robot-assisted urological surgeries, such as partial nephrectomy, radical cystectomy, and radical prostatectomy will be conducted using the Micro Hand S robot or the da Vinci robot.

Main measures: The main outcome was the success rate of operation. Surgical success was defined as that the surgical procedures were completed by the experimental or control product without transferring to non-robotic surgery. Secondary outcomes included intra- and post-operative complications, comprehensive complication index, assembly time, operation time, intraoperative hemorrhage, postoperative pain, resident time, surgeon satisfaction, incidence of adverse events, instrument malfunction, vital signs, routine blood test, hepatic and liver function.

Background:

Prostate cancer is a common disease of elderly male. With the continuous growth of life expectancy, the change of diet structure and the improvement of diagnostic technology, the incidence rate of prostate cancer has increased in recent years. Radical prostatectomy can be performed for cancer confined within the prostate capsule, which is also the best treatment for prostate cancer. At present, the commonly used surgical methods include traditional open prostatectomy, laparoscopic prostatectomy, and robot-assisted prostatectomy.

Minimally invasive surgery has always been the unremitting pursuit of surgeons. In the past decade, da Vinci robot system has expanded rapidly in China, especially in some fields of Urology, showing great advantages. In July 2000, da Vinci robotic surgery system was approved by FDA for clinical surgery. In July 2001, binder and others completed the world's first da Vinci robotic surgery system assisted laparoscopic radical prostatectomy. Since then, da Vinci robotic surgery has been widely used in clinical surgery worldwide, such as Urology, general surgery, cardiothoracic surgery, obstetrics and Gynecology, pediatric surgery, etc. In recent ten years, da Vinci robotic surgery in China has developed rapidly, and the number of urological surgery cases is increasing rapidly. It is widely used in radical prostatectomy, partial nephrectomy, radical cystectomy, pyeloplasty, adrenalectomy and other urological surgery. This is mainly due to the unique anatomical structure of Urology, which enables da Vinci system to take its advantages such as 3D high-definition vision, precise cutting and separation, intracavitary suture technology, and short learning curve.

The special anatomical position of the prostate and the surrounding anatomical structure determine the difficulty of the operation. In terms of learning curve, it needs 50-100 cases for laparoscopic surgery to pass the learning curve, and it needs 10-20 cases for da Vinci robotic surgery system to pass the learning curve; In terms of visual field, the anatomy of robot assisted surgery is clearer, which is conducive to the protection of urethral membrane and neurovascular bundle, and sexual function, and the "double construction" of anatomy and function. In addition, it also has the characteristics of less bleeding and complications, rapid postoperative recovery, short hospital stay, and can achieve the same or better oncological and functional results.

In nephrectomy or partial nephrectomy, compared with laparoscopic surgery, the learning curve is greatly shortened; By providing high-resolution and three-dimensional images, magnifying the images can make the surgical field clearer; Moreover, the da Vinci robotic surgery system has seven degrees of freedom, which can simulate the movement of the hand, so that the surgeon can better complete the incision, fine suture and reconstruction, zoom action, tremor filtering, which can alleviate the hand fatigue of the surgeon, greatly increase the safety of hand surgery, reduce the time of renal warm ischemia, and maximize the protection of renal function.

In conclusion, when performing radical prostatectomy, radical cystectomy or partial nephrectomy using robot surgery system, it has certain advantages compared with laparoscopic surgery, and it also needs to record its related complications, especially electrical machinery related complications.

Method:

The study was designed as a single-blind prospective randomized clinical trial since it is inevitable for the surgeon to know what kind of robot to use during the operation. After obtaining the approval of the Ethics Review Committee and other relevant institutions, a total of 136 patients will be included in this study from from July 2022 to November 2023 (anticipated). Those patients will be enrolled by two hospital centers and the patients will be randomly divided into the Micro Hand S surgical robot group and the da Vinci surgical robot group. All enrolled patients were fully informed and signed the informed consent. Patients were randomly assigned to each group in a 1:1 ratio, and information of the grouping and intervention measures were not available to patients. Patients of each group were matched for age, sex, body mass index (BMI), and complications to reduce confounding intervention factors. Robot-assisted partial nephrectomy, radical cystectomy, and radical prostatectomy will be conducted using the Micro Hand S robot or the da Vinci robot. The success rate of operation, assembly time, operation time, intraoperative hemorrhage, continence rate (if applicable), postoperative pain, comprehensive complication index, resident time and surgeon satisfaction were recorded.

Robot-assisted partial nephrectomy, radical cystectomy, and radical prostatectomy will be conducted using the Micro Hand S robot or the da Vinci robot. During the operation, the assembly time, intraoperative blood loss, operation time, operation success rate, and the adjacent organ and vascular injury caused by the failure of the tested system were recorded. Pain score was analyzed 24±2 hours after the surgery. The vital signs (temperature, pulse, respiration, blood pressure) were measured on the 3rd day postoperatively. Meanwhile, the routine blood test (red blood cells, white blood cells and neutrophils, platelet, hemoglobin), liver and renal function (ALT, AST, TP, ALB, GLU, TBIL, BUN, and CREA), the electrolyte (K, Na, Cl, Ca), blood sugar, and color ultrasound of liver, gallbladder, pancreas and spleen were checked. Operating surgeons filled in the satisfaction questionnaire postoperatively. Furthermore, the patients' postoperative condition changes, postoperative medication, postoperative complications, and resident time were also recorded. All the patients were followed up by telephone at 30±5 days postoperatively to evaluate the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* BMI was 18-30 kg/m2;
* patients that need partial nephrectomy, radical cystectomy, and radical prostatectomy.
* patients that understand the benefits and risks of this test, and are willing to participate and sign the informed consent form

Exclusion Criteria:

* Previous abdominal and pelvic surgery history (preoperative evaluation may affect this operation)
* People with serious uncontrolled diseases or acute infections, including but not limited to: Patients with active tuberculosis and HIV antibody positive; Those who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and whose copy number of hepatitis B virus DNA (HBV-DNA) is higher than the lower limit of detection or the range of normal values; Hepatitis C virus (HCV) antibody positive; Treponema pallidum positive patients; Covid-19 positive patients
* Long term use of anticoagulant and antiplatelet drugs (antiplatelet aggregation drugs were stopped less than 1 week before operation), and patients with a history of hemorrhagic diseases or hematopoietic dysfunction or coagulation dysfunction; Serious allergic constitution and suspected or confirmed alcohol, drug or drug addiction; Patients with epilepsy or mental history or cognitive impairment
* Patients with cardiovascular and cerebrovascular diseases, blood system diseases, or poor control of blood glucose and blood pressure, who cannot tolerate anesthesia or increase the risk of surgery according to the evaluation of the researcher
* women in pregnancy or lactation
* Patients who have participated or are participating in clinical research of other drugs, biological agents or medical devices in the past 3 months
* Other conditions that the researcher believes are not suitable to participate in this experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of the surgery | after the study is completed, up to 18 months
  the proportion of patients with successful operation in all participating patients in the experimental or control group

SECONDARY OUTCOMES:
assembly time | after the robot is assembled, all data will be collected within 18 months
  The assembly time extends from the time the robot starts to the time the trocar is connected to the robot arm.

OTHER OUTCOMES:
blood loss | after the procedure is completed, all data will be collected within 14 months
  Intraoperative blood loss is the total amount of blood loss from the beginning of the operation (after the robot was assembled) to the incision is sutured.
The hospital stay | from the admission to the discharge, all data will be collected within 14 months
  The hospital stay is the total number of days from the admission to the discharge of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No